CLINICAL TRIAL: NCT04869865
Title: The Effects of a Springtime Home Cleanse on Skin, Gut, Metabolic and Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: AyurPrana LLC (Unknown); Pearl Banyan, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYURCLN-01
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: mental health; skin health; gut health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All subjects will be given the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Detoxification cleanse
  Interventions: Dietary Supplement: 9-day detoxification cleanse and 1 week of pre-cleanse transition

INTERVENTIONS:
Dietary Supplement: 9-day detoxification cleanse and 1 week of pre-cleanse transition — Subjects will participate in the full 9-day Springtime Home Cleanse, including the week prior to a pre-cleanse transition period. The cleanse includes a transition week, 9 days of a monodiet, internal oleation with ghee, external oleation, herbs, purgation, and an enema. During this time, subjects will also attend daily online meetings on Facebook Live throughout the cleanse and on AyurPrana's AyurLearn online portal to participate in guided mediation and yoga. Subjects will also use these platforms to access daily cleanse instructions and journaling topics.

SUMMARY:
This pilot study will evaluate the effects of a Springtime Home Cleanse on skin, gut, metabolic, and mental health. The study will also assess changes in overall quality of life. The results will be used to design a larger cleanse-based study in the future.

DETAILED DESCRIPTION:
Short-term dietary cleanses and other popular detoxification methods are thought to eliminate accumulated toxins from the body and subsequently, promote health and well-being. Although previous studies have reported improvements in weight loss, blood pressure and insulin resistance with these practices, there is not enough scientific evidence to corroborate these claims. Therefore, the objective of this pilot study is to determine the effects of a short-term dietary cleanse on various parameters of skin, gut, metabolic and mental health and evaluate the aforementioned health claims.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (ages 18-69)
* Individuals must be able to read and comprehend study procedures and consent forms.
* Individuals who have baseline metabolic, gut or stress dysfunction
* Individuals must be able to minimize activity during the home cleanse for full participation and compliance.
* Individuals must be willing to reduce caffeine, sugar, alcohol, dairy and carbohydrate rich foods throughout the study.
* Individuals must be willing to have flash photo facial images taken with imaging systems.

Exclusion Criteria:

* Individuals with a known allergy to lime or lime juice, ginger or ginger pickle, turbinado sugar, rock salt, curcumin, coriander, fennel, cardamom, cinnamon, trikatu, yellow mung dal, kitchari spice, triphala, dashamula and guduchi powder, castor oil and chyavanprash.
* Individuals who are lactose intolerant, or with a known allergy to ghee.
* Individuals who are in the process of being vaccinated.
* Individual who have a history of gastrointestinal inflammatory diseases or a history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis) or other similar systemic diseases in the opinion of the investigator.
* Individuals who are recovering from a serious illness (requiring hospitalization), infection (requiring hospitalization), or surgery within one month of starting the study or unwilling to wait one month after their illness, infection, or surgery prior to starting the study.
* Individuals who are recovering from a non-serious illness or infection who are recovered and unwilling to wait 2 weeks from their illness or infection.
* Individuals who are in a concurrent intervention based clinical research study at this site or any other facility in the past two weeks.
* Has a condition or is on a medication the investigator and/or designee believes could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results.
* Individuals who have had exposure to systemic antibiotics within the month prior or unwilling to wash out for a month.
* Women who are pregnant or breastfeeding.
* Individuals who are cognitively impaired.
* Prisoners

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-29 (Estimated); Primary Completion 2022-04-03 (Estimated); Study Completion 2022-04-03 (Estimated)

PRIMARY OUTCOMES:
Microbiota diversity | 3 weeks
  Evaluation of gut microbiome diversity
Microbiome intestinal markers | 3 weeks
  Zonulin, calprotectin, antibodies against LPS

SECONDARY OUTCOMES:
Serum hemoglobin A1c (HbA1c) levels | 3 weeks
  Evaluate serum HbA1c level via ZRT Laboratories Cardiometabolic Panel
Serum high-sensitivity C-reactive protein (hsCRP) level | 3 weeks
  Evaluate serum hsCRP level via ZRT Laboratories Cardiometabolic Panel
Serum triglyceride (TG) level | 3 weeks
  Evaluate serum TG level via ZRT Laboratories Cardiometabolic Panel
Serum low density lipoprotein (LDL) level | 3 weeks
  Evaluate serum LDL level via ZRT Laboratories Cardiometabolic Panel
Serum high density lipoprotein (HDL) level | 3 weeks
  Evaluate serum HDL level via ZRT Laboratories Cardiometabolic Panel
Serum very low density lipoprotein (VLDL) level | 3 weeks
  Evaluate serum VLDL level via ZRT Laboratories Cardiometabolic Panel
Salivary diurnal cortisol pattern | 3 weeks
  Salivary diurnal cortisol pattern via ZRT Laboratories Saliva Hormone Test
Facial redness - image based | 3 weeks
  BTBP Clarity Mini 3D camera
Facial wrinkles - image based | 3 weeks
  BTBP Clarity Mini 3D camera
Facial trans-epidermal water loss (TEWL) | 3 weeks
  Vapometer, Delfin Technologies
Tongue changes - image based | 3 weeks
  Evaluate changes in tongue coating, discoloration, depressions, indentations, and cracking via iPad imaging
Quality of Life Survey Based Assessment | 3 weeks
  Self assessment using World Health Organization (WHO) Quality of Life Questionnaire
Safety assessments for GI distress | 3 weeks
  Self assessment using Digestive Questionnaire
Blood pressure | 3 weeks
Heart Rate | 3 weeks
Respiratory Rate | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No